CLINICAL TRIAL: NCT02775175
Title: The Influence of a Modified Ramadan Fasting Regimen on Health and Well-being in Healthy Muslims - a Randomised Controlled Trial
Brief Title: Influence of a Modified Ramadan Fasting on Health and Well-being in Healthy Muslims - a Randomised Controlled Trial
Acronym: Ramadan_16
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universität Duisburg-Essen (Other)
Responsible Party: Principal Investigator, Romy Lauche, Principle Investigator, Universität Duisburg-Essen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 15-6336-BO
Record Dates: First submitted 2016-05-14; First posted 2016-05-17 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2018-04

CONDITIONS: Healthy Volunteers
Keywords: Ramadan; Fasting; Nutrition; Quality of Life
MeSH Terms: conditions — Fasting

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fasting as Usual (No Intervention): This group will continue to practice their usual fasting regimen during Ramadan
- Modified Ramadan Fasting (Experimental): This group will receive an educational intervention providing knowledge about fasting and its effects on the body/mind, and health advice around nutrition to support health and well-being of participants during Ramadan.
  Interventions: Behavioral: Modified Ramadan Fasting

INTERVENTIONS:
Behavioral: Modified Ramadan Fasting — The intervention aims to provide knowledge about fasting and its effects on the body/mind, and health advice around nutrition to support health and well-being of participants during Ramadan.
  Arms: Modified Ramadan Fasting

SUMMARY:
In this study the investigators will test the impact of a modified Ramadan Fasting regimen on health and well-being. The 2016 Ramadan is around summer solstice in Germany making it one of the most challenging fasting periods for participating Muslims. The modified Ramadan Fasting consists of educational components around fasting, and advice for nutritional modifications in order to support health and well-being during Ramadan, while the control group will continue to fast as usual. The investigators will measure not only body weight/fat but also include measures of psychological well-being, and spiritual practice, and serum markers for blood lipids, and blood sugar. With this trial the investigators aim to determine, whether such modifications around Ramadan will be beneficial for health and well-being.

DETAILED DESCRIPTION:
see above

ELIGIBILITY:
Inclusion Criteria:

* Healthy Muslims participating in Ramadan Fasting
* No first time fasting

Exclusion Criteria:

* Untreated or malign hypertension
* Eating disorder
* psychological disorder (e.g. depression, schizophrenia, addiction)
* co-morbid disease (e.g. diabetes, cancer, gout)
* pregnancy
* breastfeeding women
* BMI under 20 or above 40
* recently on a diet

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 114 (Actual)
Dates: Start 2016-05; Primary Completion 2016-07 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Quality of life | 4 weeks
  Quality of life, measured by the WHO-5 (World Health Organisation, Allgaier et al., 2011, WHO-5, 1998)
  WHO-5, Fragebogen zum Wohlbefinden (Version 1998), Psychiatric Research Unit, WHO Collaborating Centre in Mental Health, http://www.who-5.org/.

SECONDARY OUTCOMES:
Quality of life | 16 weeks
  Quality of life, measured by the WHO-5 (World Health Organisation, Allgaier et al., 2011, WHO-5, 1998)
  WHO-5, Fragebogen zum Wohlbefinden (Version 1998), Psychiatric Research Unit, WHO Collaborating Centre in Mental Health, http://www.who-5.org/.
Satisfaction with life | 4 weeks
  Satisfaction with life, measured by the BMLSS-10 (Brief Multidimensional Life Satisfaction Scale)
  Büssing A, Fischer J, Haller A, Heusser P, Ostermann T, Matthiessen PF: Validation of the brief multidimensional life satisfaction scale in patients with chronic diseases. European Journal of Medicine Research 2009; 14: 171-177
Satisfaction with life | 12 weeks
  Satisfaction with life, measured by the BMLSS-10 (Brief Multidimensional Life Satisfaction Scale)
  Büssing A, Fischer J, Haller A, Heusser P, Ostermann T, Matthiessen PF: Validation of the brief multidimensional life satisfaction scale in patients with chronic diseases. European Journal of Medicine Research 2009; 14: 171-177
Spirituality | 4 weeks
  Spirituality, measured by the SpREUK-P SF17 (Spiritual and Religious Attitudes in Dealing with Illness)
  Büssing A, Reiser F, Michalsen A, Baumann K: Engagement of patients with chronic diseases in spiritual and secular forms of practice: Results with the shortened SpREUK-P SF17 Questionnaire. Integrative Medicine: A Clinician´s Journal 2012; 11(1):28-38
Spirituality | 12 weeks
  Spirituality, measured by the SpREUK-P SF17 (Spiritual and Religious Attitudes in Dealing with Illness)
  Büssing A, Reiser F, Michalsen A, Baumann K: Engagement of patients with chronic diseases in spiritual and secular forms of practice: Results with the shortened SpREUK-P SF17 Questionnaire. Integrative Medicine: A Clinician´s Journal 2012; 11(1):28-38
Sleep quality | 4 weeks
  Sleep quality, measured by the PROMIS Sleep Disturbances and Sleep-related impairment questionnaires
  Yu L, Buysse DJ, Germain A, Moul DE, Stover A, Dodds NE, Johnston KL, Pilkonis PA. Development of short forms from the PROMIS™ sleep disturbance and Sleep-Related Impairment item banks. Behav Sleep Med. 2011 Dec 28;10(1):6-24.
Sleep quality | 12 weeks
  Sleep quality, measured by the PROMIS Sleep Disturbances and Sleep-related impairment questionnaires
  Yu L, Buysse DJ, Germain A, Moul DE, Stover A, Dodds NE, Johnston KL, Pilkonis PA. Development of short forms from the PROMIS™ sleep disturbance and Sleep-Related Impairment item banks. Behav Sleep Med. 2011 Dec 28;10(1):6-24.
Mindfulness | 4 weeks
  Mindfulness, measured by the Conscious Presence and Self Control Instruments
  Büssing A, Walach H, Kohls N, Zimmermann F, Trousselard M. Conscious Presence and Self Control as a measure of situational awareness in soldiers - A validation study. International Journal of Mental Health Systems 2013, 7:1
Mindfulness | 12 weeks
  Mindfulness, measured by the Conscious Presence and Self Control Instruments
  Büssing A, Walach H, Kohls N, Zimmermann F, Trousselard M. Conscious Presence and Self Control as a measure of situational awareness in soldiers - A validation study. International Journal of Mental Health Systems 2013, 7:1
Inner Peace | 4 weeks
  Inner Peace, measured by the Functional Assessment of Chronic Illness Therapy - Spiritual Well-Being Scale (FACIT-Sp)
  Peterman AH, Fitchett G, Brady MJ, Hernandez L, Cella D: Measuring spiritual well-being in people with cancer: the functional assessment of chronic illness therapy - Spiritual Well-being Scale (FACIT-Sp). Ann Behav Med 2002, 24:49-58.
Inner Peace | 12 weeks
  Inner Peace, measured by the Functional Assessment of Chronic Illness Therapy - Spiritual Well-Being Scale (FACIT-Sp)
  Peterman AH, Fitchett G, Brady MJ, Hernandez L, Cella D: Measuring spiritual well-being in people with cancer: the functional assessment of chronic illness therapy - Spiritual Well-being Scale (FACIT-Sp). Ann Behav Med 2002, 24:49-58.
Ease of life | 4 weeks
  Ease of life, measured by the Emotional and rational disease acceptance questionnaire (ERDA)
  Büssing A, Matthiessen PF, Mundle G. Emotional and rational disease acceptance in patients with depression and alcohol addiction. BMC Health and Quality of Life Outcomes 2008; 6:4.
Ease of life | 12 weeks
  Ease of life, measured by the Emotional and rational disease acceptance questionnaire (ERDA)
  Büssing A, Matthiessen PF, Mundle G. Emotional and rational disease acceptance in patients with depression and alcohol addiction. BMC Health and Quality of Life Outcomes 2008; 6:4.
Body weight | 4 weeks
  Body weight in kg
Body weight | 12 weeks
  Body weight in kg
Body fat | 4 weeks
  Body fat, measured using a Bioelectrical impedance analysis scale
Body fat | 12 weeks
  Body fat, measured using a Bioelectrical impedance analysis scale
Waist circumference | 4 weeks
  Waist circumference in cm
Waist circumference | 12 weeks
  Waist circumference in cm
Hip circumference | 4 weeks
  Hip circumference
Hip circumference | 12 weeks
  Hip circumference
Blood pressure | 4 weeks
  Blood pressure, measured using an automatic device
Blood pressure | 12 weeks
  Blood pressure, measured using an automatic device
Heart rate | 4 weeks
  Heart rate, measured using an automatic device
Heart rate | 12 weeks
  Heart rate, measured using an automatic device
Compliance | 4 weeks
  Compliance, measured using a structured interview about nutrition during Ramadan
Adverse events | 4 weeks
  adverse events during the study period
Blood lipid level | 4 weeks
  Blood lipid level, including serum measures triglycerides, cholesterol, HDL and LDL cholesterol
Blood glucose level | 4 weeks
  Blood glucose level, serum measure
AST/SGOT | 4 weeks
  AST/SGOT, as measure of liver function
ALT/SGPT | 4 weeks
  ALT/SGPT, as measure of liver function
GGT | 4 weeks
  GGT, as measure of liver function
Uric acid level | 4 weeks
  Uric acid level, serum measure
Creatinine | 4 weeks
  Creatinine level, serum measure

CONTACTS AND LOCATIONS:
Overall Officials: Gustav Dobos, MD, Study Director — Department of Internal and Integrative Medicine, Kliniken Essen-Mitte, Faculty of Medicine, University of Duisburg-Essen
Locations (1):
- Department of Internal and Integrative Medicine, Kliniken Essen-Mitte, Essen, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lauche R, Fathi I, Saddat C, Klose P, Al-Abtah J, Büssing A, Rampp T, Dobos G, Cramer H. The effects of Ramadan fasting on physical and mental health in healthy adult Muslims - Study protocol for a randomised controlled trial. Advances in Integrative Medicine, 2016, 3 (1), 26 - 30. doi: 10.1016/j.aimed.2016.07.001
- [Derived] Lauche R, Fathi I, Saddat C, Klose P, Al-Abtah J, Bussing A, Rampp T, Dobos G, Cramer H. Effects of Modified Ramadan Fasting on Mental Well-Being and Biomarkers in Healthy Adult Muslims - A Randomised Controlled Trial. Int J Behav Med. 2024 May 22. doi: 10.1007/s12529-024-10296-0. Online ahead of print. PMID 38777939